CLINICAL TRIAL: NCT05940844
Title: A Phase 1b, Open-label, Non-randomized Trial for the Assessment of Safety, Tolerability, and Pharmacokinetics of OB-002 as a Monotherapy in Patients With Refractory Metastatic Colorectal, Pancreatic, Gastric, Breast, or Urothelial Cancer
Brief Title: Study of OB-002 in Patients With Refractory Metastatic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study terminated due to changes in the drug development plan
Sponsor: Orion Biotechnology Polska Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OB-002-101
Record Dates: First submitted 2023-06-16; First posted 2023-07-11 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Cancer; Metastatic Colorectal Cancer; Metastatic Pancreatic Cancer; Metastatic Gastric Cancer; Metastatic Breast Cancer; Metastatic Urothelial Carcinoma
Keywords: solid tumors; CCR5
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Breast Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: A total of up to 36 patients will be screened and 18 enrolled. At least 3 patients at each of the 4 dose levels (0.25, 0.5, 1.0, and 1.5 mg/kg planned) and up to 6 patients at the highest dose(s) if no MTD. An additional 3 patients may be recruited at any of the dose levels to define the dose(s) for further development. Each patient will be enrolled for at least one 28-day cycle of treatment with a FU period of up to 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- open label OB-002 monotherapy 0.25 mg/kg (Experimental): Dose Level 1
  Interventions: Drug: OB-002
- open label OB-002 monotherapy 0.5 mg/kg (Experimental): Dose Level 2
  Interventions: Drug: OB-002
- open label OB-002 monotherapy 1.0 mg/kg (Experimental): Dose Level 3
  Interventions: Drug: OB-002
- open label OB-002 monotherapy 1.5 mg/kg (Experimental): Dose Level 4
  Interventions: Drug: OB-002
- open label OB-002 monotherapy expansion cohort (Experimental): Dose Expansion
  Interventions: Drug: OB-002

INTERVENTIONS:
Drug: OB-002 — The patients will be dosed once weekly (Days 1, 8, 15 and 22) over a 4-week treatment cycle with a 28 day dose-limiting toxicity (DLT) observation period.

SUMMARY:
This is an open-label, non-randomized trial with OB-002 monotherapy dose escalation followed by a dose expansion in patients with metastatic colorectal, pancreatic, gastric, breast, or urothelial cancer who have progressed on two or more treatment regimens.

DETAILED DESCRIPTION:
The dose escalation will use a conventional 3+3 approach, at a minimum of four planned dose levels (0.25, 0.5, 1.0, and 1.5 mg/kg), to establish a maximum tolerated dose (MTD). Additional dose levels may be investigated if PK, pharmacodynamic (PD), safety, and efficacy data indicate higher dose levels may be appropriate. The first patient - sentinel patient - at each dose level will be observed for three days before additional patients can be dosed within the same dose level.

The patients will be dosed once weekly (Days 1, 8, 15, and 22) over a 4-week treatment cycle with a 28-day dose-limiting toxicity (DLT) observation period. After a full cohort has completed Day 28 assessments there will be a pause for safety evaluation conducted by the Safety Monitoring Committee (SMC). Once safety data have been reviewed, the SMC will make their recommendations to Orion who will decide whether to proceed to dosing the next dose cohort. Screening may continue during the SMC pause.

Once all patients in the highest planned cohort (1.5 mg/kg OB 002) have completed Day 28 assessments, safety, PK, receptor occupancy (RO), and tolerability data will be reviewed to determine which dose level should be expanded or whether an additional dose level is needed. The expanded cohort will enrol 6 patients at the identified dose level.

Patients may remain on treatment until disease progression with a follow-up (FU) period of up to 12 months. All adverse events (AEs) and non-invasive tumor assessments will be documented throughout the FU period to characterize the objective response rate (ORR) and, progression-free survival (PFS). Patients that do not complete the DLT observation period for non-DLT reasons will be replaced

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Patients at least 18 years of age on the day of providing consent.
3. Patients with accessible metastatic lesions for repetitive biopsy retrieval.
4. Patients with histologically or cytologically confirmed metastatic colorectal, pancreatic, gastric, breast, or urothelial tumors who have progressed or were intolerant after two or more regimens and for whom no standard of care or curative therapy options are available.
5. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 within 7 days of the start of treatment
6. Patients with evaluable and measurable lesions as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
7. Patients with adequate organ function at the time of enrollment as defined below:

   1. Neutrophil count ≥1500/mm3
   2. Platelet count ≥7.5 × 105/mm3
   3. Hemoglobin >9.0g/dL (transfusion >2 weeks before testing permitted)
   4. Aspartate transaminase (AST), alanine transaminase (ALT)

      ≤2.5 × the upper limit of normal (ULN) (≤5-times in patients with liver metastasis)
   5. Total bilirubin ≤1.5 × ULN
   6. Creatinine clearance >60 mL (determined by Cockcroft-Gault Equation)
   7. International normalized ratio (INR) ≤1.5 × ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT)
8. In women with the potential for pregnancy (including patients with amenorrhea due to medical reasons, such as chemical menopause), after consenting to the study, the patient must agree to use contraception from enrollment and for at least 12 weeks after taking the final dose of the investigational drug. Women with the potential for pregnancy include those who have begun menstruation, who have not undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy, and who have not gone through menopause. Menopause is defined as the consecutive absence of menstrual periods for ≥12 months. Total abstinence is an acceptable mode of contraception.
9. In the case of men, the patient must agree after consenting to the study to use contraception from enrollment and for at least 13 weeks after taking the final dose of the investigational drug (a period of 90 days [the spermatogenesis cycle] is added to 5-times the elimination half-time of I/O agent. Total abstinence is an acceptable mode of contraception.

Exclusion criteria:

1. Unwilling to undergo biopsy retrieval during screening (unless an archival sample taken within 3 months before screening is available) and after the fourth infusion of OB-002
2. Patients who have undergone systemic chemotherapy, radiotherapy, surgery, or hormone therapy <28 days before enrollment, also see exclusion criterion #8.

   Note: Patients must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Patients with ≤Grade 2 neuropathy may be eligible. If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
3. Patients with a history of CCR5 antagonist therapy (e.g., vicriviroc, maraviroc).
4. Patients with uncontrolled hypertension (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg) with treatment
5. QTc interval greater than 450 msec (males) or 470 msec (females)
6. Patients with acute coronary syndrome (including myocardial infarction and unstable angina), and with a history of coronary angioplasty or stent placement performed within 6 months before enrollment
7. Patients with a large amount of pleural effusion or ascites requiring more than weekly drainage
8. Patients with a history of (non-infectious) pneumonitis that required steroids or have current pneumonitis.
9. Patients with a ≥Grade 3 active infection according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
10. Patients with symptomatic brain metastasis (1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system [CNS] disease)
11. Patients with partial or complete gastrointestinal obstruction
12. Patients with interstitial lung disease requiring treatment with systemic steroids or other agents
13. Patients who test positive for either anti-human immunodeficiency virus type 1 (HIV-1) antibodies, hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (HCV) antibodies with a positive HCV RNA viral load test
14. Patients with concurrent autoimmune disease, or a history of chronic or recurrent autoimmune disease
15. Patients who require systemic corticosteroids equivalent to ≥10 mg prednisone (excluding temporary usage for tests, prophylactic administration for allergic reactions, or to alleviate swelling associated with radiotherapy) or immunosuppressants, or who have received such a therapy <14 days before enrollment in the present study
16. Patients with a history or findings of ≥Grade 3 congestive heart failure according to the New York Heart Association functional classification
17. Patients with a seizure disorder who require pharmacotherapy
18. Persistent proteinuria >3.5 g/24 hours measured by urine protein-creatinine ratio from a random urine sample (≥Grade 3, NCI CTCAE v5.0)
19. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
20. Major surgical procedure or significant traumatic injury within 28 days before the start of study medication
21. Non-healing wound, non-healing ulcer, or non-healing bone fracture
22. Patients with evidence or history of any bleeding diathesis, irrespective of severity
23. Any hemorrhage or bleeding event ≥Grade 3 (NCI CTCAE v 5.0) within 4 weeks prior to the start of the study medication
24. Women who are pregnant or breastfeeding, or with the potential for pregnancy unwilling to undergo contraception
25. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Safety: adverse events | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Number of patients experiencing adverse events (AEs), serious AEs (SAEs) abnormalities in clinical laboratory tests, vital signs, electrocardiograms (ECGs), and physical exams
Safety: Maximum Tolerated Dose | From date of first infusion with 28 days observation period (+/-3 days)
  MTD will be defined on the basis of dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
(PK) Pharmacokinetics Cmax | samples are collected from first to fourth infusion (period of 28 days +/- 2 days)
  To evaluate the multiple-dose pharmacokinetic (PK) profile of OB-002 with maximum observed concentration (Cmax) profile of OB-002 in patients with refractory metastatic colorectal, pancreatic, breast, or urothelial cancer.
(PK) Pharmacokinetics Tmax | samples are collected from first to fourth infusion (period of 28 days +/- 2 days)
  To evaluate the multiple-dose pharmacokinetic (PK) profile of OB-002 with time to maximum serum concentration (Tmax) in patients with refractory metastatic colorectal, pancreatic, breast, or urothelial cancer.
(PK) Pharmacokinetics AUC0-t | samples are collected from first to fourth infusion (period of 28 days +/- 2 days)
  To evaluate the multiple-dose pharmacokinetic (PK) profile of OB-002 with area under the curve from time 0 to last sampling time (AUC0-t) in patients with refractory metastatic colorectal, pancreatic, breast, or urothelial cancer.
(PK) Pharmacokinetics AUC0 ∞ | samples are collected from first to fourth infusion (period of 28 days +/- 2 days)
  To evaluate the multiple-dose pharmacokinetic (PK) profile of OB-002 with area under the curve from time 0 to infinity (AUC0 ∞) in patients with refractory metastatic colorectal, pancreatic, breast, or urothelial cancer.
(PK) Pharmacokinetics t1/2 | samples are collected from first to fourth infusion (period of 28 days +/- 2 days)
  To evaluate the multiple-dose pharmacokinetic (PK) profile of OB-002 with terminal half-life (t1/2) in patients with refractory metastatic colorectal, pancreatic, breast, or urothelial cancer.
(PK) Pharmacokinetics Vd | samples are collected from first to fourth infusion (period of 28 days +/- 2 days)
  To evaluate the multiple-dose pharmacokinetic (PK) profile of OB-002 with the volume of distribution (Vd) in patients with refractory metastatic colorectal, pancreatic, breast, or urothelial cancer.
(PK) Pharmacokinetics CL | samples are collected from first to fourth infusion (period of 28 days +/- 2 days)
  To evaluate the multiple-dose pharmacokinetic (PK) profile of OB-002 with clearance (CL) in patients with refractory metastatic colorectal, pancreatic, breast, or urothelial cancer.

OTHER OUTCOMES:
Exploratory: immunogenicity of OB-002 | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  A number of patients developing antidrug antibodies (ADA) and the titers developed in these participants.
Exploratory: evaluation of receptor occupancy (RO) of OB-002 in blood | samples are collected from first to fourth infusion (period of 28 days +/- 2 days)
  Percent of CCR5 receptors occupied by OB-002 in blood
Exploratory: evaluation of receptor occupancy (RO) of OB-002 in tumor | samples are collected from first to fourth infusion (period of 28 days +/- 2 days)
  Percent of CCR5 receptors occupied by OB-002 in tumor biopsies
Exploratory: preliminary efficacy of OB-002 as monotherapy based on best overall response | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months, assessed up to 12 months
  Objective response rate (ORR): defined as the proportion of patients having best overall response (BOR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by the investigator.
Exploratory: preliminary efficacy of OB-002 as monotherapy based on complete response | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months, assessed up to 12 months
  Objective response rate (ORR): defined as the proportion of patients having complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by the investigator.
Exploratory: preliminary efficacy of OB-002 as monotherapy based on partial response | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months, assessed up to 12 months
  Objective response rate (ORR): defined as the proportion of patients having a partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by the investigator.
Exploratory: preliminary efficacy of OB-002 as monotherapy based on Progression-free survival | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months, assessed up to 12 months
  Progression-free survival (PFS): defined as the time from randomization until objective tumor progression or death, whichever comes first by RECIST v1.1
Exploratory: evaluation of OB-002 on blood biomarkers (immune cells) | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Systemic monitoring of circulating immune cells
Exploratory: evaluation of OB-002 on blood biomarkers (cytokines) | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Systemic monitoring of secreted cytokines.
Exploratory: evaluation of OB-002 on blood biomarkers (chemokines) | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Systemic monitoring of secreted chemokines.
Exploratory: evaluation of OB-002 on tumor biomarkers (tumor-associated immune cells in TMI) | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Examination of tumor-associated immune cells in tumor microenvironment
Exploratory: evaluation of OB-002 on blood biomarkers (TCR) | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Genomic analyses on whole blood/peripheral blood mononuclear cells (PBMC) for T-cell repertoire (TCR) analyses
Exploratory: evaluation of OB-002 on blood biomarkers (ctDNA) | From first infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Plasma circulating tumor DNA (ctDNA) analysis

IPD SHARING:
Plan to Share IPD: No